CLINICAL TRIAL: NCT00829959
Title: Attitudes About Childbearing And Fertility In Women Seeking Genetic Testing For Inherited Breast And Ovarian Cancer Syndromes (HBOC)
Brief Title: Attitudes About Childbearing And Fertility With Inherited Breast And Ovarian Cancer Syndromes (HBOC)
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0624
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Ovary, Cancer; Ovarian Cancer; Breast Cancer; Hereditary Breast and Ovarian Cancer Syndrome; HBOC; Genetic testing; Pregnancy; Fertility; Prenatal diagnostic testing
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Genetic Counseling: Women referred to the Clinical Cancer Genetics Program for discussion of Hereditary Breast And Ovarian Syndrome (HBOC).
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — 1 - 2 questionnaires, lasting 10-15 minutes.
  Other Names: Survey

SUMMARY:
Objectives:

- To evaluate the attitudes and opinions of women undergoing genetic counseling for hereditary breast and ovarian cancer syndrome, both before and after testing, in regards to pregnancy and fertility

Hypothesis:

-Factors that will increase the percentage of women endorsing prenatal diagnostic testing will include a personal history of breast or ovarian cancer, having had a mother or sister die of breast or ovarian cancer, and testing positive for a BRCA mutation.

DETAILED DESCRIPTION:
This questionnaire is part of a study at The University of Texas M.D. Anderson Cancer Center. The purpose is to ask women who are seeking genetic testing for HBOC their viewpoints surrounding fertility, childbearing and parenting, both at the time of testing and at the time of results disclosure. The aim is to evaluate if the genetics results disclosure may influence women's views regarding these topics. Researchers hope to use this information to provide more information to the patient and the caregiver to help both parties with this very important cancer survivorship issue.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have been referred to the Clinical Cancer Genetics Program for discussion of Hereditary Breast And Ovarian Syndrome (HBOC).
2. Participants must be seen by clinical cancer geneticist and undergo genetic counseling here at M.D. Anderson Cancer Center for HBOC.
3. Participants may or may not have a personal diagnosis of cancer.
4. Participants may have already seen or undergone reproductive endocrine evaluation and had any reproductive treatment.
5. The participant must be a woman and have reproductive potential which would include either active menstruation, blood tests with premenopausal ranges of Luteinizing Hormone (LH), Follicle Stimulating Hormone (FSH) and estradiol, or was premenopausal prior to starting chemotherapy for a diagnosed breast cancer.
6. Age >/= 18 years old
7. The patient must be able to speak and read fluently in either English or in Spanish in order to complete the questionnaire.

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing genetic counseling within UT MDACC Clinical Cancer Genetics Program for hereditary breast and ovarian cancer syndrome (HBOC).
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2009-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Women Endorsing Prenatal Diagnostic Testing (Questionnaire response) | Baseline and post genetic testing (results disclosure) at 3-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Litton, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org